CLINICAL TRIAL: NCT03685552
Title: Safety Evaluation of a Diet and Nutritional Supplementation Program for Support of Balanced Bowel Function in Healthy Volunteers
Brief Title: Safety Evaluation of a Diet and Nutritional Supplementation Program- Purify 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's Sunshine Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSP-CT-012
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Gastrointestinal Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prog: Purify-2 (Experimental): All subjects will be participating in a diet life style modification program (High Phytopro dietary program) ( a modified Mediterranean style low glycemic load food plan) and will be receiving a supportive nutritional supplements over a 4 week period.
  Interventions: Other: Prog: Purify-2

INTERVENTIONS:
Other: Prog: Purify-2 — Nutritional Supplements to be administered:
  * Protein Shakes: one protein shake twice a day
  * Probiotics (Bacillus Coagulans) once a day
  * Biome NO+ ( blend of amino acids, specifically l-arginine and l-citrulline, combined with red beet root, grape polyphenol extract, vitamins and minerals) twice a day
  * In.Form Purify ( blend of psyllium hull, inulin, L-glutamine, fruit, fruit extracts and zinc) twice a day

SUMMARY:
The study evaluated the safety, tolerability and acceptability of a lifestyle modification program with nutritional supplementation designed to restore balance to healthy bowel function in generally healthy subjects

DETAILED DESCRIPTION:
To investigate the safety, tolerance and acceptability of a lifestyle modification and targeted nutraceuticals for balanced bowel function in generally healthy volunteers. To evaluate safety and tolerability, blood samples were drawn for blood counts, metabolic profiles, plasma lipids, and additional cardiovascular risk factors. Quality of life questionnaires, medical symptom questionnaire were evaluated at baseline, week 1, week 2 and week 4. Vitals signs, weight and body composition were monitored at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 and ≤ 69 years old
* Generally healthy and meeting entrance criteria
* Score ≥ 8 points on the Purify Readiness Scale (Appendix B)
* Willingness to make required lifestyle changes during study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Change in prescription medications, over-the-counter medications, medical foods, and nutritional supplements within 30 days prior to Day 1 and for the duration of the study.
* Use of medications classified as narcotics 15 days prior to Day 1 and for the duration of the study.
* Use of prescription medications and/or over-the-counter medications for acute and semi-acute medical conditions 15 days prior to Day 1 and for the duration of the study. Use of acetaminophen is permitted on an as-needed basis.
* Use of an investigational drug or participation in an investigational study within 30 days prior to Day 1 and for the duration of the study.
* Use of oral or injectable corticosteroids within 30 days prior to Day 1 and for the duration of the study.
* Use of anticoagulant medications (heparin compounds, platelet inhibitors or warfarin) within 30 days prior to Day 1 and for the duration of the study. Use of aspirin 81 mg or 325 mg once daily is permitted.
* Use of neuro-active prescription medications specifically major and atypical antipsychotic medications within 30 days prior to Day 1 and for the duration of the study.
* Use of prescription medications, over-the-counter medications, medical foods, and nutritional supplements for the treatment of hyperlipidemia within 30 days prior to Day 1 and for the duration of the study.
* Use of prescription medications, over-the-counter medications, medical foods, and nutritional supplements for the treatment of hyperglycemia within 30 days prior to Day 1 and for the duration of the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0). | 4 weeks
  Data collection at individual and group visits and physician interviews at individual visits (baseline, week 1, week 2 and week 4) will be used to assess participants for treatment-related adverse events. Subjects with ongoing AEs may be followed for an additional 4 weeks at the discretion of the PI.

SECONDARY OUTCOMES:
Changes in Quality of life questionnaire [Medical Outcomes Study-Short Form 36 (MOS-SF36)] compared to baseline | 4 weeks
  The clinician will review the Medical Outcomes Study-Short Form 36 (MOS-SF36)] at individual visits (baseline, week 1, week 2 and week 4).
Changes in gastrointestinal Quality of Life questionnaire with Bristol Stool Chart scores compared to baseline | 4 weeks
  The clinician will review the Gastrointestinal Quality of Life questionnaire with Bristol Stool Chart scores at individual visits (baseline, week 1, week 2 and week 4).
Changes in Medical Symptom Questionnaire compared to baseline | 4 weeks
  The clinician will review the Medical Symptom Questionnaire at individual visits (baseline, week 1, week 2 and week 4).
Number of participants with treatment-related changes in basic safety labs | 4 weeks
  Phlebotomy will be conducted at individual visits (baseline, week 1, week 2 and week 4).
  Comprehensive Metabolic Panels (CMP) including ALT (Alanine aminotransferase), AST(aspartate aminotransferase) and Complete Blood Counts (CBC) will be assessed for treatment-related change from baseline.
Changes in blood pressure and peripheral pulse compared to baseline | 4 weeks
  Blood pressure and peripheral pulse will be monitored at individual visits (baseline, week 1, week 2 and week 4).
Changes in weight in pounds compared to baseline | 4 weeks
  Weight in pounds will be monitored at individual visits (baseline, week 1, week 2 and week 4).
Changes in body fat in percentage compared to baseline | 4 weeks
  Body fat in percentage will be monitored at individual visits (baseline, week 1, week 2 and week 4).
Changes in body mass index (BMI) in kg/m2 compared to baseline | 4 weeks
  Body mass will be monitored at individual visits (baseline, week 1, week 2 and week 4).
Changes in waist circumference in inches compared to baseline | 4 weeks
  Body mass will be monitored at individual visits (baseline, week 1, week 2 and week 4).
Changes in lipid panel compared to baseline | 4 weeks
  Lipid panel will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in inflammatory marker (high sensitivity C-reactive protein (hs-CRP) in mg/L) to identify low levels of inflammation that can be associated with conditions like cardiovascular disease compared to baseline | 4 weeks
  hs-CRP will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Gammaglutamyl transferase (GGT) in U/L compared to baseline | 4 weeks
  GGT will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in fasting Glucose and Insulin compared to baseline | 4 weeks
  Glucose and Insulin will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in inflammatory markers levels including calprotectin, secretory Immunoglobulin A (IgA), and eosinophil-derived neurotoxin | 4 weeks
  Calprotectin, secretory IgA, and eosinophil-derived neurotoxin will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in myeloperoxidase (MPO) levels compared to baseline | 4 weeks
  MPO will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Heme Oxygenase-1 (HO-1) levels in ng/ml compared to baseline | 4 weeks
  (HO-1) will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in total branch chain amino acids levels compared to baseline | 4 weeks
  Total branch amino acids will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Trimethylamine N-oxide/ Asymmetric dimethylarginine/ Symmetric dimethylarginine (TMAO/ADMA/SDMA) levels compared to baseline | 4 weeks
  TMAO/ADMA/SDMA will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in sodium copper chlorophyllin levels compared to baseline | 4 weeks
  Chlorophyllin will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in metallothionein protein levels compared to baseline | 4 weeks
  Metallothionein will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Thiobarbituric acid (TBARS/Malondialdehyde) compared to baseline | 4 weeks
  TBARS will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Total Antioxidant Capacity (TAC) levels as Trolox Equivalent (TE) compared to baseline | 4 weeks
  TAC will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in serum Zonulin levels compared to baseline | 4 weeks
  Zonulin will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in Lactulose/Mannitol ratio in 24-hour urine collected samples compared to baseline | 4 weeks
  Lactulose/Mannitol ratio will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in urine toxic element levels compared to baseline | 4 weeks
  Toxic element levels will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in stool Zonulin levels compared to baseline | 4 weeks
  Stool Zonulin will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in stool short chain fatty acids (SCFAs) levels including n-butyrate, propionate and acetate compared to baseline | 4 weeks
  SCFAs levels will be measured at individual visits (baseline, week 1, week 2 and week 4).
Changes in stool Firmicutes count, Bacteroidetes count, and Firmicutes/Bacteroidetes ratio compared to baseline | 4 weeks
  stool Firmicutes count, Bacteroidetes count, and Firmicutes/Bacteroidetes ratio will be measured at individual visits (baseline, week 1, week 2 and week 4).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Lamb, MD, Principal Investigator — Hughes Center for Research and Innovation
Locations (1):
- The Hughes Center for Research and Innovation, Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delzenne NM, Cani PD. Interaction between obesity and the gut microbiota: relevance in nutrition. Annu Rev Nutr. 2011 Aug 21;31:15-31. doi: 10.1146/annurev-nutr-072610-145146. PMID 21568707
- [Background] de Vrese M, Schrezenmeir J. Probiotics, prebiotics, and synbiotics. Adv Biochem Eng Biotechnol. 2008;111:1-66. doi: 10.1007/10_2008_097. PMID 18461293
- [Background] Macfarlane GT, Steed H, Macfarlane S. Bacterial metabolism and health-related effects of galacto-oligosaccharides and other prebiotics. J Appl Microbiol. 2008 Feb;104(2):305-44. doi: 10.1111/j.1365-2672.2007.03520.x. PMID 18215222
- [Background] Roberfroid M, Gibson GR, Hoyles L, McCartney AL, Rastall R, Rowland I, Wolvers D, Watzl B, Szajewska H, Stahl B, Guarner F, Respondek F, Whelan K, Coxam V, Davicco MJ, Leotoing L, Wittrant Y, Delzenne NM, Cani PD, Neyrinck AM, Meheust A. Prebiotic effects: metabolic and health benefits. Br J Nutr. 2010 Aug;104 Suppl 2:S1-63. doi: 10.1017/S0007114510003363. PMID 20920376
- [Background] Lamb JJ, Konda VR, Quig DW, Desai A, Minich DM, Bouillon L, Chang JL, Hsi A, Lerman RH, Kornberg J, Bland JS, Tripp ML. A program consisting of a phytonutrient-rich medical food and an elimination diet ameliorated fibromyalgia symptoms and promoted toxic-element detoxification in a pilot trial. Altern Ther Health Med. 2011 Mar-Apr;17(2):36-44. PMID 21717823